CLINICAL TRIAL: NCT02243072
Title: Translating Home-Based Interventions for Adolescents With Poorly Controlled TID
Brief Title: Home-Based Interventions for Adolescents With Type 1 Diabetes
Acronym: R34
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Deborah Ellis, Ph.D., Professor of Family Medicine and Public Health Sciences Wayne State University School of Medicine, Wayne State University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34DK102091-01 (NIH); R34DK102091 (NIH)
Record Dates: First submitted 2014-09-04; First posted 2014-09-17 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2016-11

CONDITIONS: Type 1 Diabetes
Keywords: Insulin Dependent Diabetes Mellitus; family therapy; adolescents; regimen adherence; metabolic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fit Familes plus Standard Medical Care (Experimental): Participants will receive the intervention Fit Families plus Standard Medical Care which is an adaptation of Multisystemic Therapy for Type 1 Diabetes delivered by Community Health Workers (CHWs) in addition to standard medical care.
  Interventions: Behavioral: Fit Families plus Standard Medical Care
- Standard Medical Care (No Intervention): Standard medical care is provided at Children's Hospital of Michigan consistent with the standards for the care of children with T1D outlined by the American Diabetes Association.

INTERVENTIONS:
Behavioral: Fit Families plus Standard Medical Care — Adolescents will receive the Fit Families plus Standard Medical Care which consists of twice weekly home-based, family psychotherapy from a CHW for 6 months
  Arms: Fit Familes plus Standard Medical Care

SUMMARY:
Adolescents with T1D and chronic poor metabolic control are at high risk for short and long-term diabetes complications and are heavy users of both medical resources and health care dollars. The purpose of the proposed study is to collaborate with a community agency to develop and test an intervention, Fit Families, that uses the core components of a previously successful home-based family treatment, but that can delivered by lower cost community health workers. If successful, Fit Families could improve health outcomes in a vulnerable population at high risk for diabetes complications, and could be translated to real-world treatment settings.

DETAILED DESCRIPTION:
The proposed study is a planning grant in which MST will be adapted for delivery by community health workers and will be conducted in collaboration with CHASS, a community agency providing health care to underserved residents of Detroit with diabetes. The new intervention, Fit Families (FF), will be tested in a pilot randomized controlled trial in order to evaluate FF feasibility, finalize outcome measures, estimate intervention effect sizes on health outcomes (i.e., youth adherence, glycemic control, quality of life) and determine potential cost savings associated with reduced hospital admissions. These steps will allow for finalization of intervention content and other trial parameters in preparation for a larger R18 dissemination trial.

The design for the proposed study is a randomized, controlled trial using a sample of 60 adolescents. Half will be randomly assigned to the treatment intervention, Fit Families plus standard medical care, and the other half will be assigned to standard medical care alone. Families who are randomized to FF receive intensive, home-based family therapy delivered by a community health worker (CHW) for approximately six months.

ELIGIBILITY:
Inclusion Criteria:

* a current hemoglobin A1c(HbA1c) of >9.0%
* an average HbA1c of >9.0% during the past year
* reside in the metro Detroit tri-county area
* diagnosed with Type 1 diabetes for at least one year
* aged 10-17
* patient of Children's Hospital of Michigan Diabetes Clinic

Exclusion Criteria:

* severe mental impairment/thought disorder
* Active suicidality
* Active homicidality
* Diabetes secondary to another comorbid medical condition and/or medical management differing substantially from that of most children with diabetes.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Metabolic Control: Hemoglobin A1c (HbA1c) | Change from Baseline at 7 months, Change from Baseline at 9 months
  retrospective measure of blood glucose control, encompasses the previous 2-3 months

SECONDARY OUTCOMES:
DKA admissions and emergency room (ER) Visits: hospital information systems data extraction, Service Utilization Questionnaire (SUQ) | Change from Baseline at 7 months, Change from Baseline at 9 months
  The number of patient visits to acute care settings represents a significant health care cost in this high-risk population.
Quality of life | Change from Baseline at 7 months, Change from Baseline at 9 months
  44 scale item designed to tap life satisfaction, diabetes impact and diabetes related worries in adolescents.
Regimen Adherence: Diabetes Management Scale (DMS), Glucose Meter Downloads | Change from Baseline at 7 months, Change from Baseline at 9 months
  The DMS assesses a broad range of management behaviors, such as insulin management, dietary management, blood glucose monitoring, symptom response, and parent assistance/supervision. Glucose meters only assess blood glucose monitoring, but are empirically linked to metabolic control

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Ellis, Ph.D, Principal Investigator — Wayne State University
Locations (1):
- Children's Hospital of Michigan, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No